CLINICAL TRIAL: NCT04792632
Title: Clinical Performance Evaluation of Veye Lung Nodules
Acronym: CPEVLN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aidence (Industry)
Responsible Party: Sponsor
Other Study IDs: Aidence01
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Lung; Node

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Intervention: Intervention is the use of Veye Lung Nodules during the reading of the CT scans
  Interventions: Device: Veye Lung nodules

INTERVENTIONS:
Device: Veye Lung nodules — Veye Lung Nodules

SUMMARY:
Veye Lung Nodules (Aidence B.V., Amsterdam, the Netherlands) is a medical software device that is intended to assist radiologists with pulmonary nodule management on CT chest scans.

This clinical trial aims to assess the clinical performance of Veye Lung nodules via a standalone performance evaluation and a reader study.

ELIGIBILITY:
Inclusion Criteria:

- Subjects that underwent a CT chest scan for either lung cancer screening or routine practice

Exclusion Criteria:

* Subjects with >10 pulmonary nodules;
* Subjects with pulmonary mass(es) = largest axial diameter >30mm;
* Subjects with interstitial lung disease.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: US adult population that received a CT chest scan either as part of a lung cancer screening program or during routine practice
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Detection accuracy | 2 months
  Demonstrate that the accuracy for detecting actionable pulmonary nodules by radiologists using the device (AIDED) is superior to that of radiologists not using the device (UNAIDED)

SECONDARY OUTCOMES:
Segmentation accuracy | 1 month
  Demonstrate that the accuracy for segmenting actionable pulmonary nodules by the device is non-inferior to expert radiologists

OTHER OUTCOMES:
Growth assessment accuracy | 1 month
  Demonstrate that the accuracy for determining volume change of actionable pulmonary nodules by the device is non-inferior to expert radiologists
Composition classification accuracy | 2 months
  Demonstrate that the accuracy for classifying the composition of actionable pulmonary nodules by radiologists using the device (AIDED) is superior to that of radiologists not using the device (UNAIDED)

CONTACTS AND LOCATIONS:
Locations (1):
- Intrinsic Imaging, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No